CLINICAL TRIAL: NCT01131741
Title: Comparison of Perfusion Index, T Wave Amplitude, Systolic Blood Pressure and Heart Rate as an Indicator for Detecting Intravascular Injection of Epinephrine Containing Test Dose During Operation in Anesthetized Adults
Brief Title: Comparison of Perfusion Index, T Wave Amplitude, Systolic Blood Pressure and Heart Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jin Huh, MD., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-2009-141
Record Dates: First submitted 2010-05-23; First posted 2010-05-27 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Injections, Intravenous
Keywords: anesthesia, general; blood pressure; epinephrine; heart rate; injections, intravenous
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epinephrine (Experimental)
  Interventions: Drug: Epinephrine
- Control (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Epinephrine — This group receives 3 mL of 1% lidocaine containing epinephrine IV during operation.
  Arms: Epinephrine
Drug: Control — This group receives 3 mL of saline IV during operation.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether changes in perfusion index can be used for detecting intravascular injection of an epinephrine in anesthetized adults and to compare its reliability with criteria using changes in heart rate, systolic blood pressure or T-wave amplitude.

DETAILED DESCRIPTION:
Intravenous injection of local anesthetics could result in life-threatening complications during general anesthesia. Physicians usually use local anesthetics containing epinephrine to detect intravascular injection. Existing methods including heart rate, systolic blood pressure and T-wave amplitude are unreliable to detect intravascular injection during anesthesia and a method using changes in perfusion index was recently suggested. This study was designed to determine whether perfusion index is a reliable method to detect intravascular injection of epinephrine containing local anesthetics and to compare its reliability with conventional criteria in sevoflurane anesthetized adults.

We will randomize patients to 2 groups: a saline group and an epinephrine group. Changes in perfusion index, systolic blood pressure, heart rate and T-wave amplitude will be measured during 5 minutes after injection of 3 mL of saline or 1% lidocaine containing epinephrine. we will determine sensitivity, specificity, positive predictive value and negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 patients undergoing general anesthesia for elective surgery

Exclusion Criteria:

* emergent operation
* those who are taking anticoagulant medication, calcium channel blockers, or b-blockers
* laparoscopic operation
* history of smoking

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
change of perfusion index from baseline | during 5 min after injection of epinephrine containing test dose or saline
  we will observe the change of perfusion index from baseline during 5 min after injection of epinephrine containing test dose or saline. Patients whose perfusion index decrease more than 25% are defined as positive response.we will obtain the sensitivity, specificity, positive predictive value, negative predictive value using perfusion index criteria to determine the reliability of perfusion index criteria.

SECONDARY OUTCOMES:
change of systolic blood pressure, heart rate, T-wave amplitude from baseline | during 5 min after injection of epinephrine containing test dose or saline

CONTACTS AND LOCATIONS:
Overall Officials: Jin Huh, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea